CLINICAL TRIAL: NCT06868017
Title: Randomized Controlled Clinical Study of Efficacy and Safety of Initumab Combined with Pyrrotinib and Chemotherapeutic Agents in Neoadjuvant Therapy for HER2-positive Breast Cancer with Different Treatment Cycles
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-206
Record Dates: First submitted 2025-02-18; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: HER2 Positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Queue A (Other)
  Interventions: Drug: Cohort A will receive an initial load dose of 8mg/kg and a maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 4 doses
- Queue B (Other)
  Interventions: Drug: Cohort B will receive an initial load dose of 8mg/kg and a maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 6 doses

INTERVENTIONS:
Drug: Cohort A will receive an initial load dose of 8mg/kg and a maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 4 doses — Cohort A will receive initumab at initial load dose of 8mg/kg and maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 4 doses. Pyrrotinib 400mg orally once daily; Combined chemotherapy drugs (not limited, according to the actual clinical selection), a total of 4 cycles of administration
  Arms: Queue A
Drug: Cohort B will receive an initial load dose of 8mg/kg and a maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 6 doses — The initial loading dose of initumab was 8mg/kg, and the maintenance dose was 6mg/kg, which was administered intravenously on the first day of every three weeks. Pyrrotinib 400mg orally once daily; Combined chemotherapy drugs (not limited, according to the actual clinical selection), a total of 6 cycles of administration
  Arms: Queue B

SUMMARY:
The purpose of this study was to explore the efficacy and safety of initumab combined with pyrrotinib and chemotherapy for 4 cycles and 6 cycles of neoadjuvant therapy for HER2-positive breast cancer, and to explore the efficacy and safety of continued use of initumab combined with pyrrotinib in pCR patients.

This study adopted A prospective, randomized controlled, open-label design, and selected eligible subjects to be randomly divided into cohort A and Cohort B. Cohort A will receive initumab at initial load dose of 8mg/kg and maintenance dose of 6mg/kg intravenously on the first day of every three weeks for a total of 4 doses. Pyrrotinib 400mg orally once daily; Combined chemotherapy drugs (not limited, according to the actual clinical selection), a total of 4 cycles of administration. After surgery for breast cancer, initumab + pyrrotinib was selected as adjuvant therapy for pCR patients after surgery for 1 year (neoadjuvant therapy + adjuvant therapy for a total of 1 year, a total of 13 cycles of adjuvant therapy), and non-pCR patients were selected by doctors. Cohort B will receive initumab at initial load dose of 8mg/kg and maintenance dose of 6mg/kg intravenously on the first day of every three weeks. Pyrrotinib 400mg orally once daily; Combined chemotherapy drugs (not limited, according to the actual clinical selection), a total of 6 cycles of administration. After surgery for breast cancer, initumab + pyrrotinib was selected as adjuvant therapy for pCR patients after surgery for 1 year (neoadjuvant therapy + adjuvant therapy for a total of 1 year, and adjuvant therapy for a total of 11 cycles), and non-pCR patients were selected by doctors.

ELIGIBILITY:
inclusion criteria：

1. Age ≥18 years old, while ≤70 years old, gender is not limited; 2.2. Invasive breast cancer confirmed histologically by air-core needle biopsy; According to AJCC breast cancer Staging System 8th edition, clinical staging was T1c-4, N0-3, M0.

3. HER2 positive: IHC 3+ or IHC 2+ and FISH+ 4.Left ventricular ejection fraction (LVEF) ≥ 50% 5.ECOG physical condition score is 0 or 1 6.In the absence of blood transfusion or symptomatic treatment (granulocyte colony-stimulating factor/erythropoietin (EPO)/interleukin-11, etc.) within 14 days prior to initial administration, organ function must meet the following requirements Blood routine: absolute value of neutrophil (ANC) ≥1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin (Hb) ≥90g/L Blood biochemistry: Total bilirubin (TBIL) ≤1.5×ULN; ALT and AST≤1.5×ULN; BUN and Cr≤1.5×ULN; Creatinine clearance ≥50mL/min (Cockcroft-Gault formula) 7.Voluntarily participate in this study, sign informed consent, have good compliance and are willing to cooperate with follow-up

exclusion criteria:

1. Previous history of invasive breast cancer
2. Bilateral breast cancer, inflammatory breast cancer (e.g., erythema and/or skin involvement, and/or pathological findings of tumor cells in the dermal lymphatic vessels), or clinical stage T1c, N0, M0
3. Prior biopsy of primary tumor and/or axillary lymph node excision and/or excision
4. Previous systemic treatment for breast cancer;
5. A history of life-threatening hypersensitivity, or a known history of allergy to any component of the investigational drug;
6. Participated in clinical trials of other drugs or medical devices within 4 weeks before the first drug use, and received treatment with experimental drugs or devices
7. Patients who had undergone major surgery within 28 days prior to the first dose or planned to undergo major surgery during the study period
8. Other malignant tumors (excluding cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ) within the previous 5 years
9. Active hepatitis, active tuberculosis or other serious infectious diseases, including but not limited to: Active hepatitis C virus (HCV) infection (HCV antibody positive but not RNA negative), or hepatitis B virus (HBV) infection (HBV surface antigen positive and HBV-DNA copy number >2000 IU/mL) or other serious infections requiring systemic treatment such as bacteremia, severe infectious pneumonia
10. A history of immunodeficiency or other autoimmune diseases, including but not limited to human immunodeficiency virus (HIV) infection (HIV-positive), systemic lupus erythematosus, rheumatoid arthritis, or a history of organ transplantation
11. Patients with a history of cardiovascular and cerebrovascular diseases, including: (1) unstable angina pectoris; (2) medically treatable or clinically significant arrhythmias; (3) myocardial infarction occurring within 6 months; (4) Heart failure, degree II and above atrioventricular block; (5) Cerebral infarction (except lacunar cerebral infarction), cerebral hemorrhage and other diseases occurring within 6 months
12. Patients with poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg under regular medication), or with a prior history of hypertensive crisis or hypertensive encephalopathy
13. Pregnant and lactating female patients; Pregnant women of childbearing age who were positive in screening pregnancy test; Patients who are unwilling to use effective contraception throughout the trial period and for 6 months after the end of medication
14. Other circumstances deemed inappropriate by the investigator to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-02-19 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
total Pathological Complete Response，tpCR | After completion of neoadjuvant therapy, subjects' completely removed breast specimens and all sampled regional lymph nodes were evaluated

SECONDARY OUTCOMES:
Overall Response Rate，ORR | It refers to the percentage of cases that achieved complete response (CR) and partial response (PR) after neoadjuvant therapy as a percentage of the total number of evaluable cases
Event-Free Survival，EFS | Refers to the time from enrollment to the first recorded recurrence of disease, disease progression, or death from any cause after surgery
Invasive Disease-Free Survival，iDFS | Refers to the time from enrollment to the first occurrence of an aggressive ipsilateral tumor recurrence, aggressive countermeasure breast cancer, local/regional aggressive recurrence, distant recurrence, or death from any cause
Overall Survival | Refers to the time from enrollment to death

IPD SHARING:
Plan to Share IPD: No